CLINICAL TRIAL: NCT06852937
Title: Pilot Study of Single-Port Robot-Assisted Surgery Using Da Vinci SP Surgical System for Patients With Complex Cholelithiasis and Choledocholithiasis
Brief Title: Using da Vinci SP System for Patients With Cholelithiasis and Choledocholithiasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202409006DIPD
Record Dates: First submitted 2024-12-17; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-12

CONDITIONS: Cholelithiasis; Choledocholithiasis
MeSH Terms: conditions — Cholelithiasis; Choledocholithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Operation of focus procedure with da Vinci SP Surgery System (Experimental): Operation of cholecystectomy and common bile duct exploration with da Vinci SP Surgery System
  Interventions: Device: da Vinci SP Surgery System

INTERVENTIONS:
Device: da Vinci SP Surgery System — da Vinci SP Surgery System

SUMMARY:
A prospective, interventional, single arm study to investigate clinical feasibility of single-stage cholecystectomy and common bile duct exploration using da Vinci SP Surgical System (robotic surgery)

DETAILED DESCRIPTION:
Cholelithiasis (gallstones) is a common disease of digestive tract in adults. It has been reported that 5-10% or 2 million of Taiwanese adults have gallstones according to National Health Insurance Administration.

Laparoscopic cholecystectomy is deemed a surgical standard of care for its safety, effectiveness, and benefits: less post-operative pain, faster recovery, shorter hospital stay, and better cosmesis. However, the advantages of da Vinci surgical system include enhanced vision, wristed instruments, and dexterity of control.

Robotic cholecystectomy by single-port SP system is associated with shorter operation time, shorter dissection time, and less post-operative pain.

Further improvement in robotic cholecystectomy with CBDE regarding cosmesis and patient satisfaction could be made by adopting da Vinci SP system which preserves enhanced vision and instrument dexterity with only one access port. So far there is no published data on robotic cholecystectomy with CBDE using da Vinci SP. Current study is set forth to evaluate technical feasibility and clinical outcome of robotic biliary surgery using da Vinci SP Surgical System for patients with complex cholelithiasis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 years or more
2. Symptomatic cholelithiasis with or without choledocholithiasis, symptomatic chronic cholecystitis with or without biliary tract injury or stricture
3. Indication of cholecystectomy with or without common bile duct exploration and deemed feasible for robotic surgery
4. Patient not feasible or have failed stone extraction or intervention for choledocholithiasis by endoscopic retrograde cholangiopancreatography for patients with choledocholithiasis could be included
5. ASA physical status classification 1-2 and adequate organ function
6. Patients willing and able to comply with study protocol requirements and follow-up
7. Patients who are taking anti-platelet or anti-coagulation medications are eligible for this trial, but the associated agents should be discontinued 5 days prior to the operation day. Patients who are taking Wafarin should be admitted two days earlier for bridging to Heparin. Other medications for underlying diseases can be taken as usual.
8. With informed consent

Exclusion Criteria:

1. Severe acute cholecystitis
2. Suspected biliary tract cancer or untreated biliary tract cancer
3. BMI ≥35 or BMI <18.5
4. Unable to tolerate robotic surgery position
5. Severe adhesion due to prior abdominopelvic surgery
6. Prior major upper abdominal surgery judged by the investigator as not feasible for robotic surgery
7. Active infectious disease
8. Severe concomitant illness that drastically shortens life expectancy or increases risk of therapeutic interventions, such as: severe heart disease (NYHA functional class III-IV) or severe lung disease (GOLD Group C-D)
9. Cannot follow trial-required procedures
10. Concomitant systemic or pelvic disease that increases the risk of surgery
11. Patients with coagulopathy
12. Emergency surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-12-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of conversion rate | During Surgery
  The primary performance endpoint will be assessed as the ability to successfully completed the planned procedure with da Vinci SP System, with no conversion to alternative surgery including open surgery or laparoscopy.

SECONDARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events | up to 6 months
  The safety endpoint will be assessed as the incidence of all intra-operatvie and post-operative adverse events that occur through the follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Ming Wu, Principal Investigator — Vice Superintendent of NTUCC
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No